CLINICAL TRIAL: NCT06018116
Title: A Canadian Phase II, Placebo-controlled Randomized Trial of Bicalutamide in Patients Receiving Maintenance Avelumab for Metastatic Urothelial Cancer.
Brief Title: A Canadian Trial of Bicalutamide in Patients Receiving Maintenance Avelumab for Metastatic Urothelial Cancer.
Acronym: CANUCK-01
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Results of EV302 study do not make it feasible to complete a study in second line avelumab immunotherapy. The new standard of care make this study not pertinent.
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Cancer Research Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MP-20-2024-6963
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Metastatic Urothelial Carcinoma
Keywords: bicalutamide; avelumab
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — bicalutamide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bicalutamide (Experimental): standard of care (SOC) avelumab with 150mg daily oral bicalutamide
  Interventions: Drug: Bicalutamide 150 mg
- Placebo (Placebo Comparator): standard of care (SOC) avelumab with daily oral placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bicalutamide 150 mg — nonsteroidal antiandrogen
  Other Names: standard of care avelumab
  Arms: Bicalutamide
Drug: Placebo — placebo
  Other Names: standard of care avelumab
  Arms: Placebo

SUMMARY:
This is a Phase II, multi-center, placebo-controlled randomized controlled trial of standard of care (SOC) avelumab versus SOC avelumab with bicalutamide for patients with metastatic or locally advanced urothelial carcinoma.

DETAILED DESCRIPTION:
Urothelial carcinoma (UC) is the second most common urological cancer after prostate cancer. Non-muscle invasive bladder cancer (NMIBC) is the most common form (~75%). Muscle-invasive bladder cancer (MIBC) is found at presentation in ~25% of patients, with 10-20% of NMIBC eventually becoming MIBC. Risk groups for NMIBC are based on number of tumours, stage and size. Almost half of patients with MIBC eventually progress to metastatic disease.

Treatments for metastatic urothelial carcinoma (mUC) have evolved rapidly over the last several years. Pembrolizumab demonstrated benefit as second line therapy for locally advanced and metastatic UC. Subsequently, the landmark Phase III randomized JAVELIN trial showed that the addition of avelumab as maintenance therapy following a response to chemotherapy for mUC significantly prolonged overall survival relative to best supportive care (hazard ratio (HR) = 0.69; 95% confidence interval (CI), 0.56-0.86; P = 0.001). Overall survival and progression-free survival were 21.4 months (18.9 to 26.1) and 5.5 (4.2 to 7.2) months, respectively. This trial established avelumab as the SOC treatment and initial immunotherapy for mUC following chemotherapy.

The investigators have selected a double-blind placebo-controlled randomized study design to be able to assess the pragmatic endpoint of investigator-assessed clinical progression. Randomization will assign patients 2:1 to bicalutamide 150mg daily plus SOC avelumab or placebo plus SOC avelumab. Patients will be followed every 3 months after avelumab treatment has started and until progression.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or greater and able to provide informed consent for the trial;
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 at screening;
3. Patients with histologically confirmed urothelial carcinoma;
4. Patients is a candidate for a course of maintenance avelumab treatment for metastatic or locally advanced urothelial carcinoma;
5. Male patients with partners of child-bearing potential must agree to 2 acceptable forms of birth control and be continued for at least 130 days after study drug is discontinued.

Exclusion Criteria:

1. Patients with a history of liver disease whose hepatic enzymes, alkaline phosphatase or bilirubin are greater than twice the upper limit of normal will be ineligible.
2. Patients with neutrophils (< 1,000/μL) will be ineligible.
3. Patients on androgen replacement therapy, or those with prostate cancer or other diseases currently treated with systemic hormonal therapy will be ineligible for study enrollment. Patients receiving 5-alpha reductase inhibitors will not be excluded.
4. Patients who have a concurrent malignancy other than UC within the past years for which treatment is planned within the next 6 months.
5. Patients taking an investigational drug within 2 weeks of enrollment into this study.
6. Patients receiving or planning to receive coumadin therapy.
7. Female patients with childbearing potential are excluded due to known teratogenic effects of bicalutamide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Rate of bladder tumor recurrence | 30 months
  The primary outcome will be to the time to investigator-assessed progression on avelumab therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Toren, MD, PhD, FRCSC, Study Chair — CHU de Québec - Université Laval
Locations (1):
- CHU de Québec - Université Laval, Québec, Canada

IPD SHARING:
Plan to Share IPD: No